CLINICAL TRIAL: NCT05703230
Title: Is a Preoperative Multidisciplinary Team Meeting (Cost) Effective in Optimizing Noncardiac Surgical Patient Management: The PREPARATION Study
Brief Title: Effects of Preoperative Multidisciplinary Team Meetings for High-risk, Adult, Noncardiac Surgical Patients
Acronym: PREPARATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam UMC (Other); University of Twente (Other); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-1983
Record Dates: First submitted 2022-11-04; First posted 2023-01-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Interdisciplinary Communication; Postoperative Complications; Noncardiac Surgery; Surgical Procedures, Operative; Preoperative Care; Patient Care Team; Cost-Benefit Analysis; Comorbidities and Coexisting Conditions
Keywords: multidisciplinary team meeting; preoperative; high risk surgical patients
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: cross-sectional stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative care as usual (No Intervention): Patients undergoing preoperative care as usual, which does not include a structured preoperative multidisciplinary team meeting (no sMDT meeting)
- Structured preoperative multidisciplinary team meeting (Active Comparator): Patients are discussed preoperatively in a structured preoperative multidisciplinary team meeting
  Interventions: Other: Structured preoperative multidisciplinary team meeting

INTERVENTIONS:
Other: Structured preoperative multidisciplinary team meeting — The intervention to be investigated is the introduction of a preoperative structured multidisciplinary team (sMDT) meeting for high risk noncardiac surgical patients, which is attended by at least the treating surgical specialist, an anesthesiologist and another medical consultant with expertise relevant for the patients comorbidities and preferences. In the preoperative sMDT meeting, at least the following questions will be discussed as recommended by the Dutch Perioperative Guideline:
  * Is the proposed surgical intervention appropriate care for the patient?
  * Is the risk/benefit ratio of the proposed surgical intervention acceptable for the patient?
  * Should the patient's condition be optimized before undergoing the proposed surgical intervention?
  Arms: Structured preoperative multidisciplinary team meeting

SUMMARY:
The current multicenter stepped wedge randomized cluster trial study aims to assess whether implementation of preoperative multidisciplinary team (MDT) discussions is (cost)effective for high risk noncardiac surgical patients.

The main questions to answer are:

* Primary question: Does implementation of preoperative multidisciplinary team discussions for high risk noncardiac surgical patients diminish serious adverse events as compared to care as usual at six months postoperatively or six months after multidisciplinary team discussion in case of nonsurgical treatment?
* Secondary questions: Does implementation of preoperative multidisciplinary team discussion for high risk noncardiac surgical patients improve disability, survival, functional outcome, quality of life and cost-effectiveness as compared to care as usual at six months postoperatively or six months after multidisciplinary team discussion in case of nonsurgical treatment?

Participants will be asked to answer questionnaires at baseline, 3, 6,9 and 12 months postoperatively or post MDT discussion.

Patients for whom no structured preoperative multidisciplinary discussion is installed yet (care as usual) will be compared with patients for whom a structured preoperative multidisciplinary discussion is performed (intervention).

The study will be performed in hospitals that have no established preoperative MDT meeting at the start of the study.

DETAILED DESCRIPTION:
Due to the increase in life expectancy and improved care for patients suffering from a chronic disease, the number of complex patients requiring a surgical intervention is increasing. It is important to balance the potential benefits of this surgical treatment against the risk of permanent loss of functional capacity and quality of life due to complications. European and US guidelines on perioperative care all recommend preoperative multidisciplinary team meetings for high-risk noncardiac surgical patients. However, the evidence underlying a benefit of a preoperative MDT meeting is absent and recommendations are based on expert opinion. Moreover, considerable practice variation is currently present.

This study will assess the efficacy of implementation of a preoperative structured multidisciplinary team (sMDT) meeting to optimize perioperative management for high risk noncardiac surgical patients.

The hypothesis is that implementation of preoperative sMDT meetings for high risk noncardiac surgical patients results in less serious adverse events, is more cost-effective, and improves quality of life and functional outcome at six months, compared to preoperative care as usual (control).

A preoperative structured Multidisciplinary Team (sMDT) meeting for high risk noncardiac surgical patients will be implemented in each participating center (n=14) throughout the study. In the sMDT meeting, patients' treatment plan and alternatives will be discussed by the anesthesiologist, surgical specialist and other relevant consultants or (specialized) nurses.

The primary outcome is Serious adverse events (SAEs) according to the Clavien Dindo classification grade 3 or more, at 6 months following surgery or following the preoperative sMDT meeting in case of nonsurgical management. Secondary outcomes are: functional outcome (12-item WHO Disability Assessment Schedule), survival, quality of life (WHOQOL BREF), patients' regret (including interview at 6 months), societal costs (iMCQ and iPCQ, Electronic Medical Record (EMR) data, EQ5D-5L), alterations in perioperative management and sMDT performance (MDT-MOT), and facilitators and barriers (using structured interviews health care professionals). Most secondary outcomes will be assessed at baseline, 30 days, 3, 6 and 12 months.

Subgroup analyses will take place for e.g. age groups (approximate quintiles), patient sex, size of hospital, intent of surgery, BMI categories (underweight, normal, overweight, obese, ≥super obese), ASA physical status, frailty, MET score, smoking behavior, alcohol use, comorbidity index score, planned postoperative destination, educational attainment, and employment status.

For detailed description, see below.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; and
* American Society of Anesthesiology Physical Status (ASA-PS) score is 3 or more; and
* Clinical Frailty Scale score is 4 or more; and
* Patient is planned for elective or semi-elective noncardiac surgery; and
* As stated by the Dutch perioperative guideline:
* Doubt by the surgeon or anesthesiologist (or other discipline) regarding harm-benefit ratio of the surgical procedure; or
* Doubt if the correct measures were taken to limit the perioperative risk as much as possible; or
* Doubt if the patient agrees with the surgery or the anesthesiologic treatment and expected risks.

Exclusion Criteria:

* no informed consent
* unable to communicate with patient (either directly or through third party)
* emergency surgery
* Proposed surgical intervention for which a structured preoperative multidisciplinary team meeting, similar to the current study intervention, already exists in this respective hospital at the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) | 6 months
  Serious adverse events (SAEs), defined as:
  1. Grade 3 or more on the Clavien Dindo classification following surgical intervention, or
  2. non-operative SAEs will be graded accordingly i.e., events necessitating hospital admission, surgical intervention, single or multi-organ failure, or death.

SECONDARY OUTCOMES:
Disability status | 12 months
  The disability status of the patient, measured by the 12-item WHO disability Assessment Schedule 2.0 (WHODAS 2.0). The WHODAS 2.0 results in a metric ranging from 0 to 100 ( where 0 = no disability; 100 = full disability).
Patient experienced quality of life | 12 months
  Quality of life of the patient assessed by the abbreviated World Health Organization Quality of Life (WHOQOL BREF). The WHOQOL BREF results in a percentage of 0 to 100. The higher the percentage (to 100), the better the quality of life of the participant.
Regret of decision | 12 months
  Patients regret of decision measured by a modification of the Decision Regret Scale at 3, 6 and 12 months and qualitative interviews with several patients at 6 months.
  The decision regret scale is a 5-item questionnaire, scoring statements 1 (strongly agree) to 5 (strongly disagree). Final scoring consists of reversing the scores of the two negatively phrased items, then taking the mean of the five items. Last, the mean is converted to a score ranging from 0 to 100 by subtracting 1 and multiplying by 25. A higher score may indicate greater patient regret about their made treatment decisions. The scale was modified by adding a question asking by whom the decision was made. This question is not part of the previously described scoring of the 5-item decision regret scale.
Societal costs measured by a patient cost questionnaire | 12 months
  Societal costs as measured by a cost questionnaire at baseline, 3 and 12 months, including items of the iMTA (Institute for Medical Technology Assessment) Medical Consumption Questionnaire (iMCQ) and iMTA Productivity Cost Questionnaire (iPCQ) with a recall period of 3 months.
Hospital costs as a component of societal costs | 12 months
  Hospital costs based on electronic medical record (EMR) patient data, as a component of societal costs. Measured at baseline (hospital costs over a period of 3 months prior to preoperative screening) and measured during 12 months follow up.
Quality-adjusted life years as a component of societal costs | 12 months
  Quality-adjusted life years (QALYs) measured by the EQ-5D-5L at baseline, 3 and 12 months, as a component of societal costs.
Patients' desired outcome | baseline
  Patients' desired outcome will be assessed using the Outcome Prioritization Tool (OPT) at baseline (pre-operative assessment).
Survival | 30 days, 6 months, and 1 year postoperatively
  Survival at 30 days, 6 months, and 1 year postoperatively
Adverse events | 30 days, 6 months, and 1 year postoperatively
  Adverse events at 30 days, 6 months, and 1 year postoperatively
Surgical Outcome Risk Tool (SORT) | baseline
  Calculating an estimate of the patients' risk of death within 30 days of an operation.
Revised Cardiac Risk Index for Pre-Operative Risk (RCRI) | baseline
  The RCRI estimates patients' risk of cardiac complications after noncardiac surgery. The index is constructed by 6 items. The 6 items are scored yes (+1) or no (0), adding up to a minimum score of 0 and a maximum score of 6. The score is categorised into 4 categories (0, 1, 2, ≥3) and converted to "risk of major cardiac event (95% CI)" defined as death, myocardial infarction, or cardiac arrest at 30 days after noncardiac surgery.
American College of Surgeons Surgical Risk Calculator (ACS-NSQIP (American College of Surgeons National Surgical Quality Improvement Program)) | baseline
  Estimates patients' risk of postoperative complications.
Clinical Frailty Scale (CFS) | baseline
  A judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Metabolic Equivalent of Task (MET) | baseline
  Reflecting the amount of energy used by the body during physical activity.
The number of alterations in perioperative management decided by the sMDT. | baseline
  The number of alterations in perioperative management decided by the sMDT (19, 20). Examples for alterations are (but not limited to) changes in; type of anaesthesia, type of surgery, planned postoperative intensive care admission, cancellation of surgery, additional medication or diagnostics.
The nature of alterations in perioperative management decided by the sMDT. | baseline
  The nature of alterations in perioperative management decided by the sMDT (19, 20). Examples for alterations are (but not limited to) changes in; type of anaesthesia, type of surgery, planned postoperative intensive care admission, cancellation of surgery, additional medication or diagnostics.
The number of different medical specialties invited to participate in the sMDT meeting | baseline
  The number of different medical specialties present during the sMDT meeting in order to describe the multidisciplinary attendance of the sMDT meetings.
The number of different medical specialties present during the sMDT meeting | baseline
  The number of different medical specialties present during the sMDT meeting in order to describe the multidisciplinary attendance of the sMDT meetings.
The function of attending professionals at the sMDT meeting. | baseline
  The function of attending professionals at the sMDT meeting in order to describe the multidisciplinary attendance of the sMDT meetings.
Number of sMDT discussions per site | through study completion, 3 years
  Number of sMDT discussions per site

OTHER OUTCOMES:
Performance of sMDTs using an MDT-Meeting Observational Tool (MDT-MOT) | 6 months
  In a subset of patients: Performance of sMDTs using an MDT-Meeting Observational Tool (MDT-MOT).(21) In the MDT-MOT 10 observable teamwork domains are rated on a 5-point rating scale, using descriptive anchors for the extremes and midpoint of the scale. A score of '5' represents optimal effectiveness, calibrated against recommendations within 'The Characteristics of an Effective MDT' (by the National Cancer Action Team). A score of '3' represents effectiveness that exhibits some degree of agreement with the optimum, but not consistently, and a score of '1' represents no or little agreement with the defined optimum. Scores of '2' and '4' are included in the tool but not defined to allow observers the freedom to gradate their assessment.
Facilitators and barriers to organize preoperative sMDT meetings | 6 months
  Facilitators and barriers to organize preoperative sMDT meetings are evaluated using structured interviews with health care professionals from all different medical specialties.

CONTACTS AND LOCATIONS:
Overall Officials: Nick J. Koning, MD PhD DESA, Principal Investigator — Rijnstate Hospital; Jacqueline E. Vernooij, MD, MA, Study Director — Rijnstate Hospital
Locations (14):
- Netherlands (14):
  - Stichting Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Stichting Meander Medisch Centrum, Amersfoort
  - Stichting OLVG, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Stichting Albert Schweitzer Ziekenhuis, Dordrecht
  - Groene Hart Ziekenhuis, Gouda
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Stichting Nijmeegs Interconfessioneel Ziekenhuis Canisius Wilhelmina, Nijmegen
  - Stichting Bravis Ziekenhuis, Roosendaal
  - Stichting Protestants Christelijk Ziekenhuis Ikazia, Rotterdam
  - Maxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam

IPD SHARING:
Plan to Share IPD: Yes
Data will be made accessible on request after agreement has been received from the entire project group. The principal investigator will communicate data availability with researchers sending the requests.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 12 months after publication
Access Criteria: Data will be made accessible on request after agreement has been received from the entire project group.

REFERENCES:
- [Derived] Vernooij JEM, Hobrink E, Boerlage RM, van Beest P, van de Calseijde S, Holl T, Janssen LMJ, Klinkert L, Marsman M, Nouwen MJ, Wefers Bettink MA, Preckel B, Kalkman CJ, van Leeuwen B, Festen S, Koning NJ. Characteristics and outcome of preoperative multidisciplinary team discussions for high-risk noncardiac surgical patients in the Netherlands: a multicentre prospective observational study. Br J Anaesth. 2025 Aug;135(2):449-458. doi: 10.1016/j.bja.2025.05.004. Epub 2025 Jun 6. PMID 40480911
- [Derived] Vernooij JEM, Boerlage RM, Doggen CJM, Preckel B, Dirksen CD, van Leeuwen BL, Spruit RJ, Festen S, van der Wal-Huisman H, van Basten JP, Kalkman CJ, Koning NJ; PREPARATION study investigators. Is a preoperative multidisciplinary team meeting (cost)effective to improve outcome for high-risk adult patients undergoing noncardiac surgery: the PREPARATION study-a multicenter stepped-wedge cluster randomized trial. Trials. 2023 Oct 11;24(1):660. doi: 10.1186/s13063-023-07685-3. PMID 37821994